CLINICAL TRIAL: NCT00002990
Title: Comparative Study of Intravesical BCG Standard Dose Long-Term Maintenance Versus BCG 1/3 Dose Long-Term Maintenance Versus BCG Standard Dose Short-Term Maintenance Versus BCG 1/3 Dose Short-Term Maintenance in Intermediate and High Risk Ta, T1 Papillary Carcinoma of the Urinary Bladder
Brief Title: Surgery and BCG in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30962; EORTC-30962
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine

INTERVENTIONS:
Biological: BCG vaccine

SUMMARY:
RATIONALE: Biological therapies such as BCG use different ways to stimulate the immune system and stop cancer cells from growing.

PURPOSE: This randomized phase III trial is studying four different regimens of BCG and comparing how well they work in treating patients who have undergone surgery for bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Demonstrate that after complete transurethral resection of all papillary tumors, one third dose BCG (Bacillus Calmette-Guerin vaccine; OncoTICE) is equivalent to full dose BCG and short term maintenance is equivalent to long term maintenance with respect to duration of disease free interval, recurrence rate, percentage of patients with an increase in T-category to greater than T1, and the incidence of carcinoma in situ during follow-up.
* Demonstrate that one third dose BCG and short term maintenance are associated with fewer local and systemic side effects.

OUTLINE: This is a prospective randomized study.

At 7-15 days after transurethral resection, patients will begin receiving one of the following four regimens:

* Regimen 1: One third dose Bacillus Calmette-Guerin (BCG) vaccine plus short term maintenance. Patients receive a one third dose of BCG instilled once a week for 6 weeks, followed by three weekly instillations at months 3, 6, and 12.
* Regimen 2: Full dose BCG plus short term maintenance. Patients receive a full dose of BCG instilled once a week for 6 weeks, followed by three weekly instillations at months 3, 6, and 12.
* Regimen 3: One third dose BCG plus long term maintenance. Patients receive a one third dose of BCG instilled once a week for 6 weeks, followed by three weekly instillations at months 3, 6, 12, 18, 24, 30 and 36.
* Regimen 4: Full dose BCG plus long term maintenance. Patients receive a full dose of BCG instilled once a week for 6 weeks, followed by three weekly instillations at months 3, 6, 12, 18, 24, 30, and 36.

The patient is followed every 3 months for the first 3 years, and every 6 months thereafter.

PROJECTED ACCRUAL: 1288 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the bladder of the following types:

  * Multiple (not greater than 10), resectable, T1 or Ta, grade G1-G3
  * Solitary T1 GIII tumor

PATIENT CHARACTERISTICS:

Age:

* 85 and under

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Values used to evaluate function may not exceed two times the upper limit of normal

Renal:

* Values used to evaluate function may not exceed two times the upper limit of normal

Other:

* No second malignancy except basal cell skin carcinoma
* Not pregnant or nursing
* No uncontrollable urinary tract infection
* No active tuberculosis
* No HIV antibody
* No leukemia
* No Hodgkin's disease
* No transplant recipients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior treatment with BCG

Chemotherapy:

* No cytostatic agents within the past 3 months

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1288 (Estimated)
Dates: Start 1997-03; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Dose equivalency with respect to duration of disease free interval, recurrence rate, percentage of patients with an increase in T-category to greater than T1, and the incidence of carcinoma in situ during follow-up
Dose equivalency in terms of fewer local and systemic side effects

CONTACTS AND LOCATIONS:
Overall Officials: A. P.M. Van Der Meijden, MD, PhD, Study Chair — Jeroen Bosch Ziekenhuis
Locations (40):
- Kaiser Franz Josef Hospital, Vienna, Austria
- Belgium (7):
  - Onze Lieve Vrouw Ziekenhuis Aalst, Aalst
  - Institut Jules Bordet, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Virga Jesse Hospital, Hasselt
  - AZ Groeninge - Oncologisch Centrum, Kortrijk
- France (2):
  - Hopital Edouard Herriot, Lyon
  - Hopitaux Universitaire de Strasbourg, Strasbourg
- Greece (2):
  - G. Hatzikosta General Hospital, Ioannina
  - University of Patras Medical School, Rio Patras
- Rabin Medical Center - Beilinson Campus, Petah Tikva, Israel
- Italy (8):
  - Ospedale Di Desio, Milan
  - Istituto Scientifico H. San Raffaele, Milan
  - Azienda Ospedaliera Maggiore Della Carita, Novara
  - Azienda Ospedale S. Luigi - Universita Di Turin, Orbassano, (Torino)
  - Universita Di Palermo, Palermo
  - Universita Degli Studi Di Pisa, Pisa
  - Azienda Sanitaria Ospedale San Giovanni Battista Molinette di Torino, Turin
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (10):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Amphia Ziekenhuis - locatie Langendijk, Breda
  - Leiden University Medical Center, Leiden
  - Rijnland Ziekenhuis, Leiderdorp
  - Academisch Ziekenhuis Maastricht, Maastricht
  - University Medical Center Nijmegen, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - St. Franciscus Gasthuis, Rotterdam
- Hospital Desterro, Amadora, Portugal
- Institute of Oncology - Bucarest, Bucharest, Romania
- Turkey (Türkiye) (3):
  - Marmara University Hospital, Istanbul
  - Dokuz Eylul University School of Medicine, Izmir
  - Celal Bayar University, Manisa
- United Kingdom (4):
  - St. James's University Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Freeman Hospital, Newcastle upon Tyne, England
  - Pontefract General Infirmary, Pontefract West Yorkshire, England
  - Gartnavel General Hospital, Glasgow, Scotland

REFERENCES:
- [Derived] Cambier S, Sylvester RJ, Collette L, Gontero P, Brausi MA, van Andel G, Kirkels WJ, Silva FC, Oosterlinck W, Prescott S, Kirkali Z, Powell PH, de Reijke TM, Turkeri L, Collette S, Oddens J. EORTC Nomograms and Risk Groups for Predicting Recurrence, Progression, and Disease-specific and Overall Survival in Non-Muscle-invasive Stage Ta-T1 Urothelial Bladder Cancer Patients Treated with 1-3 Years of Maintenance Bacillus Calmette-Guerin. Eur Urol. 2016 Jan;69(1):60-9. doi: 10.1016/j.eururo.2015.06.045. Epub 2015 Jul 23. PMID 26210894
- [Derived] Brausi M, Oddens J, Sylvester R, Bono A, van de Beek C, van Andel G, Gontero P, Turkeri L, Marreaud S, Collette S, Oosterlinck W. Side effects of Bacillus Calmette-Guerin (BCG) in the treatment of intermediate- and high-risk Ta, T1 papillary carcinoma of the bladder: results of the EORTC genito-urinary cancers group randomised phase 3 study comparing one-third dose with full dose and 1 year with 3 years of maintenance BCG. Eur Urol. 2014 Jan;65(1):69-76. doi: 10.1016/j.eururo.2013.07.021. Epub 2013 Jul 24. PMID 23910233
- [Derived] Oddens J, Brausi M, Sylvester R, Bono A, van de Beek C, van Andel G, Gontero P, Hoeltl W, Turkeri L, Marreaud S, Collette S, Oosterlinck W. Final results of an EORTC-GU cancers group randomized study of maintenance bacillus Calmette-Guerin in intermediate- and high-risk Ta, T1 papillary carcinoma of the urinary bladder: one-third dose versus full dose and 1 year versus 3 years of maintenance. Eur Urol. 2013 Mar;63(3):462-72. doi: 10.1016/j.eururo.2012.10.039. Epub 2012 Nov 2. PMID 23141049